CLINICAL TRIAL: NCT04939337
Title: Study to Assess the Safety and Efficacy of Allogeneic Umbilical Cord-derived Mesenchymal Stem Cells(TH-SC01), for Treatment of Complex Perianal Fistulas in Perianal Crohn's Disease.
Brief Title: A Study of TH-SC01 for Treating Complex Perianal Fistula in Perianal Crohn's Disease.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jinling Hospital, China (Other)
Collaborators: Jiangsu Topcel-KH Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Fangyu Wang, Chief of digestive department, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20181231
Record Dates: First submitted 2021-06-10; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Crohn's Disease
Keywords: Complex Perianal Fistulas
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TH-SC01 (Experimental): TH-SC01 24 mL suspension of 120 million cells as a perilesional injection, once on Day 0.
  Interventions: Drug: TH-SC01

INTERVENTIONS:
Drug: TH-SC01 — Allogeneic Umbilical Cord-derived Mesenchymal Stem cells perilesional injection. Human TH-SC01 cell injection (human umbilical cord mesenchymal stem cells for injection, 5 million cells / ml, 6.0-10.0ml / bottle)

SUMMARY:
The purpose of this study is to asses the efficacy and Safety of Allogeneic Umbilical Cord-derived Mesenchymal Stem Cells in the Treatment of Complex Perianal Fistula in Perianal Crohn's Disease.

DETAILED DESCRIPTION:
Crohn´s disease (CD) can affect any part of the digestive system and symptoms of this chronic illness include abdominal pain, bloating, nausea, vomiting and diarrhea. CD also causes bowel wall ulcers, strictures and fistulas (abnormal passages from the intestines to another organ or the skin).

There is an unmet need for effective medical therapy in CD patients with perianal fistulas, not responding to the conventional strategies, including biological therapies. The current study is designed to assess the safety and efficacy of Allogeneic Umbilical Cord-derived Mesenchymal Stem cells from healthy donors for the treatment of perianal fistulas in patients presenting CD.

Primary objective: To assess the safety (incidence of treatment emergent adverse-events) of TH-SC01

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed Informed Consent；
* 2. According to the Diagnostic Criterion for Crohn's Disease in China's 《Consensus on the Diagnosis and Treatment of Inflammatory Bowel Disease》 (2018, Beijing), Crohn's disease was diagnosed at least 6 months before the screening period；
* 3. Crohn's disease activity index (CDAI) score of 220 or less is defined as inactive or mildly active luminal Crohn's disease；
* 4. Through clinical evaluation, MRI evaluation for anal fistula patients；
* 5. Age 18 ~ 70, male or female；
* 6. The serum or urine pregnancy test of a woman of reproductive age must be negative. Both men and women must agree to use a contraceptive method；
* 7. According to the history and related examination, the general health condition is good；
* 8. The eligible patients must at least meet one of the following conditions: patients who have failed to respond to any conventional treatment, such as conventional antibiotic therapy, immunomodulatory drug therapy, anti-tumor necrosis factor (TNF) α monoclonal antibody therapy, and 5-aminosalicylic acid

Exclusion Criteria:

* 1. CDAI > 220, or due to Crohn's disease activity, treatment needs to be upgraded immediately；
* 2. Patients with abdominal and pelvic abscess or fistula diameter more than 2 cm；
* 3. Patients with rectal and/or anal stenosis and/or active proctitis (due to limited surgical procedures)；
* 4. The number of internal and / or external openings of anal fistula was more than 2 and 3 respectively;
* 5. Patients who received steroid therapy within the first 4 weeks were screened；
* 6. Abnormal laboratory test results： Liver function: total bilirubin ≥1.5 times the upper limit of normal value, aspartate aminotransferase (AST) or alanine aminotransferase (ALT)≥2.5 times the upper limit of normal value; Renal function: Creatinine clearance below 60mL/min or 1.5 times the upper normal limit of serum creatinine (measured value or calculated by the Cockcroft-Gault formula)；
* 7.Patients with malignancy or a history of malignancy, including fistula cancer of any type；
* 8. Patients with severe, progressive, uncontrollable diseases of the liver, blood, gastrointestinal (except Crohn's disease), endocrine, lung, heart, neurological, psychiatric, or brain；
* 9. HIV, syphilis antibody positive, HCV / HBV positive, tuberculosis in the infectious period, etc;
* 10. Patients who are allergic to human serum albumin, human platelet lysates, anesthetic agents or contrast agents；
* 11. Patients with contraindications to MRI scanning；
* 12. Pregnant or lactating women and subjects who cannot commit to using effective contraceptives during the trial and for 6 months after the end of the trial；
* 13. Patients who have undergone major surgery or severe trauma in the past six months；
* 14. Patients who had received any study drug within a certain period of time prior to screening；
* 15.Patients deemed ineligible to participate in this clinical trial by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Combined Remission | 24 weeks
  Combined remission is defined as the closure of all treated external openings that were draining at baseline despite gentle finger compression, and absence of abscess(es) >2 cm (in at least 2 dimensions) of the treated perianal fistula(s) confirmed by central magnetic resonance imaging (MRI) assessment or transrectal ultrasonography(TRUS)

SECONDARY OUTCOMES:
Percentage of Participants who Achieve Clinical Remission | Up to Week 24
  Clinical remission is defined as the closure of all treated external openings that were draining at baseline despite gentle finger compression.
Percentage of Participants who Achieve Clinical Response | Up to Week 24
  Clinical response is defined as closure of at least 50% of all treated external openings that were draining at baseline despite gentle finger compression.
Percentage of Participants who decrease in PDAI | 0、4、8、16、24 weeks
  PDAI is a scoring system for assessing the severity of perianal lesions associated with Crohn's disease.It consists of the following five items :(a) perianal secretions;(b) Pain and movement;(c) Sexual life;(d) Perianal manifestations;(e) Sclerosing.Each item is rated on a five-point scale from asymptomatic (0) to severe (4), with an overall score of 0 to 20.The higher the score, the more severe the disease.
Percentage of Participants who decrease in IBDQ | 0、4、8、16、24 weeks
  IBDQ questionnaire score is used to investigate the quality of life of patients. There are 32 questions in total, and each question has 1 to 7 answers of different degrees, with 1 representing the most severe degree and 7 representing the least severe degree
Percentage of Participants who decrease in VAS scale | 0、4、8、16、24 weeks
  VAS scale was used to evaluate the pain. 0 points indicated no pain, less than 3 points indicated mild pain, 4-6 points indicated pain affecting sleep but tolerable, 7-10 points indicated pain and discomfort, affecting appetite and sleep. The higher number, the pain was more obvious.
Percentage of Participants who decrease in Wexner incontinence score | 0、4weeks
  Wexner incontinence score

CONTACTS AND LOCATIONS:
Overall Officials: Wei Juan, doctor, Principal Investigator — Jinling Hospital, China
Locations (1):
- Jinling hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thoreson R, Cullen JJ. Pathophysiology of inflammatory bowel disease: an overview. Surg Clin North Am. 2007 Jun;87(3):575-85. doi: 10.1016/j.suc.2007.03.001. PMID 17560413
- [Derived] Wei J, Zhang Y, Chen C, Feng X, Yang Z, Feng J, Jiang Q, Fu J, Xuan J, Gao H, Liao L, Wang F. Efficacy and safety of allogeneic umbilical cord-derived mesenchymal stem cells for the treatment of complex perianal fistula in Crohn's disease: a pilot study. Stem Cell Res Ther. 2023 Oct 31;14(1):311. doi: 10.1186/s13287-023-03531-0. PMID 37904247
- See also: Thoreson R, Cullen JJ. Pathophysiology of inflammatory bowel disease: an overview. Surg Clin North Am. 2007 Jun;87(3):575-85. Review. — https://pubmed.ncbi.nlm.nih.gov/17560413/